CLINICAL TRIAL: NCT00340821
Title: A Study of Familial and Genetic Aspects of Adult T-Cell Leukemia/Lymphoma, Tropical Spastic Paraparesis and Infective Dermatitis in Jamaica
Brief Title: A Study of Familial and Genetic Aspects of Adult T-Cell: Leukemia/Lymphoma , Tropical Spastic Paraparesis, and Infective Dermatitis
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999996018; OH96-C-N018
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-03-01

CONDITIONS: HTLV-I
Keywords: HTLV-I

SUMMARY:
Doctors of the University of West Indies, the Caribbean Epidemiology Center (CAREC) and the National Cancer Institute have been studying the epidemiology of HTLV-I and its role in the etiology and pathogenesis of adult T-cell leukemia/lymphoma (ALT), and aggressive T-cell lymphoma. The purpose of the current study is to evaluate familial and genetic aspects of ATL and its relationship to two other HTLV-I related conditions, HTLV-I associated myelopathy also known as tropical spastic paraparesis (HAM/TSP), and infective dermatitis. Enrollment of infective dermatitis cases was recently added and the disease entity is thought to be a harbinger for later development of either ATL or HAM/TSP. The purpose of this study is to interview patients with these conditions and perform laboratory studies (specifically, HLA and other viral or genetic studies) to better understand these diseases and their relationship to the HTLV-1 virus and the family history and genetic factors that may be involved as well.

DETAILED DESCRIPTION:
Doctors of the University of West Indies, the Caribbean Epidemiology Center (CAREC) and the National Cancer Institute have been studying the epidemiology of HTLV-I and its role in the etiology and pathogenesis of adult T-cell leukemia/lymphoma (ALT), and aggressive T-cell lymphoma. The purpose of the current study is to evaluate familial and genetic aspects of ATL and its relationship to two other HTLV-I related conditions, HTLV-I associated myelopathy also known as tropical spastic paraparesis (HAM/TSP), and infective dermatitis. Enrollment of infective dermatitis cases was recently added and the disease entity is thought to be a harbinger for later development of either ATL or HAM/TSP. The purpose of this study is to interview patients with these conditions and perform laboratory studies (specifically, HLA and other viral or genetic studies) to better understand these diseases and their relationship to the HTLV-1 virus and the family history and genetic factors that may be involved as well.

ELIGIBILITY:
* INCLUSION CRITERIA:

All cases of ATL and TSP which satisfy the case definitions above. Cases will be selected regardless of HTLV-1 sero-status.

EXCLUSION CRITERIA:

Cases who have none of the first three priority family members available i.e. parents, offspring and siblings, will be excluded from this study however summary data will be maintained.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 1993-05-17; Study Completion 2011-03-01

CONTACTS AND LOCATIONS:
Locations (1):
- University of the West Indies, Kingston, Jamaica

REFERENCES:
- [Background] Rodgers-Johnson P, Gajdusek DC, Morgan OS, Zaninovic V, Sarin PS, Graham DS. HTLV-I and HTLV-III antibodies and tropical spastic paraparesis. Lancet. 1985 Nov 30;2(8466):1247-8. doi: 10.1016/s0140-6736(85)90778-0. No abstract available. PMID 2866324
- [Background] Murphy EL, Hanchard B, Figueroa JP, Gibbs WN, Lofters WS, Campbell M, Goedert JJ, Blattner WA. Modelling the risk of adult T-cell leukemia/lymphoma in persons infected with human T-lymphotropic virus type I. Int J Cancer. 1989 Feb 15;43(2):250-3. doi: 10.1002/ijc.2910430214. PMID 2917802
- [Background] Kajiyama W, Kashiwagi S, Ikematsu H, Hayashi J, Nomura H, Okochi K. Intrafamilial transmission of adult T cell leukemia virus. J Infect Dis. 1986 Nov;154(5):851-7. doi: 10.1093/infdis/154.5.851. PMID 2877031